CLINICAL TRIAL: NCT07105826
Title: Effect of Carbonated Prebiotic Beverages Versus Caloric and Non-caloric Beverages on Satiety, Glucose, Insulin, and GLP-1 Response in Healthy Male Participants
Brief Title: Impact of Prebiotic Sodas on Satiety and Metabolic Responses in Healthy Men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Elisa Marroquin, Assistant Professor, Texas Christian University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: TCU Prebiotic Sodas Study
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Olipop; Poppi; Coca Cola - Classic; Diet Coke
Keywords: Olipop; Poppi; Diet Coke; Coca Cola; GLP-1; Insulin; soda
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: The study is a prospective, interventional study, meaning it involves actively administering interventions (in this case, beverages) to participants and measuring their effects over time.
  The study employs a randomized crossover model, where each participant receives all four interventions (Olipop, Poppi, Diet Coke, and Coca-Cola Classic) in a randomized order across multiple visits. This design allows each participant to serve as their own control, reducing variability due to individual differences and increasing statistical power with a smaller sample size.
  The study is single-blind, meaning participants are unaware of which beverage they are consuming during each visit. Beverages are served in unlabeled black containers to minimize bias in their perception of satiety, taste, or metabolic responses.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prebiotic Soda 1 (Experimental): Olipop is a low-calorie, carbonated prebiotic beverage (~20-35 kcal per 355 mL serving).
  Interventions: Other: Prebiotic Soda 1
- Prebiotic Soda 2 (Experimental): Poppi is a low-calorie, carbonated prebiotic beverage (~20-35 kcal per 355 mL serving).
  Interventions: Other: Prebiotic Soda 2
- Diet Coke (Experimental): Diet Coke is a non-caloric, carbonated beverage sweetened with artificial sweeteners. It contains zero calories and zero sugar
  Interventions: Other: Diet Soda
- Coca Cola (Experimental): Coca Cola is a caloric carbonated beverage containing high fructose corn syrup as its primary sweetener. It is considered to be a high-caloric drink (140 kcal per 355 mL serving) with 39 g of sugar.
  Interventions: Other: Regular Coke

INTERVENTIONS:
Other: Prebiotic Soda 1 — A single dose of 12 ounces of Olipop will be provided to the 10 participants while fasted. Blood samples will be collected at baseline (before the drink) and at 15, 30, 60, 90, and 120 minutes after the drink.
  Arms: Prebiotic Soda 1
Other: Prebiotic Soda 2 — A single dose of 12 ounces of Poppi will be provided to the 10 participants while fasted. Blood samples will be collected at baseline (before the drink) and at 15, 30, 60, 90, and 120 minutes after the drink.
  Arms: Prebiotic Soda 2
Other: Diet Soda — A single dose of 12 ounces of Diet Coke will be provided to the 10 participants while fasted. Blood samples will be collected at baseline (before the drink) and at 15, 30, 60, 90, and 120 minutes after the drink.
  Arms: Diet Coke
Other: Regular Coke — A single dose of 12 ounces of Regular Coke will be provided to the 10 participants while fasted. Blood samples will be collected at baseline (before the drink) and at 15, 30, 60, 90, and 120 minutes after the drink.
  Arms: Coca Cola

SUMMARY:
The study aims to study healthy men aged 18-40 to explore how different beverages affect hunger, blood sugar, insulin, and a hormone called GLP-1, which helps regulate appetite and blood sugar. The tested beverages include two prebiotic sodas (Olipop and Poppi), Diet Coke, and Coca-Cola Classic.

What's the study about? It aims to understand how these drinks influence how full participants feel and how the body handles sugar and hormones compared to each other. This could help us learn more about how prebiotic drinks, which may support gut health, compare to regular sugary or diet sodas.

What will participants do?

Participants will visit our lab at TCU (Rickel Building, rooms 256/259) four times over four weeks, with each visit lasting about 2-2.5 hours. Participants will need to fast for 8-12 hours before each visit. Here's what happens:

* First visit involves participants' consent, measurement of height and weight, and performing a finger-stick test to check blood sugar and HbA1C. Participants will also fill out questionnaires about health, diet, and beverage preferences.
* Visits 2-4: In visit 2, a DEXA scan will be performed to assess body composition. In visits 2-4, participants will drink one of the four beverages (in a random order, served in an unlabeled black container to prevent drink identification). Other variables measured at these time points include blood pressure, fasting glucose, insulin, and GLP-1. Participants will also complete questionnaires about hunger and how the drink tastes.

Each visit is spaced out by a week, and the total time commitment is about 10.5 hours. The study is expected to complete participant recruitment by December 10, 2025.

Who can join? Ten healthy men aged 18-40 who don't have diabetes, heart disease, kidney or liver issues, or other specific health conditions. Participants shouldn't smoke, vape, or have certain dietary habits like intermittent fasting. Participants will be screened to confirm eligibility.

What are the risks? The risks are low but include discomfort from blood draws or the IV catheter, a small chance of infection, and minimal radiation exposure from the DEXA scan (similar to everyday background radiation). There's also a small risk of a data breach, but participant information will be secured with password-protected systems and use ID numbers instead of names.

What do participants get? Participants will receive a DEXA scan, baseline blood sugar, and HbA1C tests. If participants have abnormal results (like high blood sugar), doctor visits would be recommended. There are no direct benefits to participants, but participation could help develop better dietary recommendations in the future.

How is privacy protected? Data will be stored securely on password-protected computers and in locked lab facilities, following HIPAA rules. Blood samples will be frozen for up to 10 years for possible future research (with participants' consent) and labeled with an ID number, not participants' names.

How to join? Participants will be recruited through flyers, emails, social media, and TCU classes. If interested, participants will complete an online screening form or scan a QR code on our flyer. If eligible, participants will be contacted to confirm details and explain the study further.

If participants have questions or want to join, contact Dr. Elisa Marroquin at e.marroquin@tcu.edu or Matthew Loritz at m.loritz@tcu.edu. Participation is voluntary, and participants can withdraw at any time, though data will be kept for analysis.

DETAILED DESCRIPTION:
Study Overview This research study, conducted by the Texas Christian University (TCU) Department of Nutritional Sciences and Kinesiology, aims to investigate the effects of carbonated prebiotic beverages (Olipop and Poppi) compared to caloric (Coca-Cola Original) and non-caloric (Diet Coke) beverages on satiety, blood glucose, insulin, and glucagon-like peptide-1 (GLP-1) responses in healthy male participants aged 18-40. The study is a single-blind, randomized crossover trial designed to explore how these beverages influence metabolic and appetite-related outcomes, addressing gaps in understanding the physiological impacts of functional beverages containing prebiotics versus widely consumed caloric and non-caloric alternatives.

Objectives and Hypotheses The primary objective is to evaluate the acute effects of four beverages-Olipop, Poppi, Diet Coke, and Coca-Cola Classic-on satiety, plasma glucose, insulin, and GLP-1 levels. Secondary objectives include assessing body composition and beverage palatability and gastrointestinal (GI) symptoms. The hypothesis is that prebiotic beverages will enhance satiety and GLP-1 secretion due to fiber content, potentially via gut microbiota fermentation, without significantly increasing glucose or insulin levels compared to Coca-Cola. Diet Coke may elicit a modest GLP-1 and satiety response due to artificial sweeteners, but minimal glucose/insulin changes. Coca-Cola is expected to cause significant glucose and insulin spikes due to its high sugar content. Additionally, hunger is expected to be reduced across all conditions, with prebiotic beverages potentially showing superior satiety effects.

Study Design

* Type: Prospective, interventional, single-blind, randomized crossover trial.
* Participants: 10 healthy males aged 18-40, accounting for a 30% attrition rate.
* Duration: Four visits, each 2-2.5 hours, separated by a one-week washout period (total ~10.5 hours).
* Randomization and Blinding: Each participant consumes all four beverages in random order, served in unlabeled black containers to minimize bias.
* Data Collection: Anthropometric measurements, body composition (DEXA scan), biochemical markers (glucose, insulin, GLP-1), and survey data (satiety, GI symptoms, beverage preference) are collected.

Study Procedures

1. Screening and Visit 1:

   * Informed consent is obtained, followed by measurement of height, weight, and blood pressure.
   * A finger-stick test assesses fasting blood glucose and HbA1c.
   * Participants complete demographic, health, beverage preference, and 3-day food log questionnaires.
2. Visits 2-4:

   * A DEXA scan measures body composition (visit 2 only).
   * Participants fast for 8-12 hours before each visit.
   * Blood pressure is measured, and fasting status is confirmed via finger-stick.
   * An intravenous catheter is inserted for blood sampling at 0, 15, 30, 60, 90, and 120 minutes post-beverage consumption to measure glucose, insulin, and GLP-1.
   * Participants consume one beverage (355 mL) within 5 minutes.
   * Satiety Questionnaires are completed at baseline and specific intervals.
   * GI Symptomps Questionnaire are filled out 24h after each visit.
   * Beverage Rating QUesitonnaire will be applied at the end of each visit.
   * Total blood volume per visit is approximately 30 mL.

Beverages Tested

* Olipop and Poppi: Prebiotic sodas containing inulin and other fibers, low calories (~20-35 kcal).
* Diet Coke: Non-caloric, sweetened with aspartame (46 mg).
* Coca-Cola Original: Caloric (140 kcal, 39 g of sugar).

Recruitment and Screening

* Methods: Flyers, emails, social media, and in-person recruitment in TCU classes.
* Process: Potential participants complete an online screening form by following the QR code from the flyers and emails. Eligible candidates undergo phone screening to confirm inclusion/exclusion criteria and receive a study overview.

Data Collection and Analysis

- Anthropometric, body composition, biochemical, and survey data will be collected as indicated in Outcome Measures.

Risks and Mitigation

1. Blood Draw/IV Catheter: Low risk of discomfort, bruising, or infection; mitigated by trained personnel and sterile techniques.
2. DEXA Scan: Minimal radiation exposure (~0.1 mSv, equivalent to background radiation); limited to one scan.
3. Data Breach: Risk minimized by deidentification, secure storage, and restricted access to IRB-approved personnel.
4. GI Discomfort: Possible with prebiotic beverages; monitored via GI Symptoms Questionnaire.

Benefits

* Direct: Participants receive a $150 gift card, DEXA scan results, baseline glucose, and HbA1c levels (finger sticks)
* Indirect: No direct benefits, but results may inform evidence-based recommendations for beverage consumption.

Results Sharing

* Baseline finger-stick results (glucose, HbA1c, lipids) are shared at testing.
* Lab-measured glucose and insulin levels, analyzed in batches after all participants complete the study, will not be shared, as delayed analysis limits immediate clinical utility.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male
* Age: 18-40 years
* Health Status: Healthy, with no significant medical conditions
* Body Mass Index (BMI): 18.5-24.9 kg/m²

Exclusion Criteria

* Diabetes: Diagnosed diabetes (Type 1 or Type 2)
* Gastrointestinal Disorders: Any diagnosed gastrointestinal conditions (e.g., irritable bowel syndrome, inflammatory bowel disease)
* Liver Disease: Any diagnosed liver conditions
* Kidney Disease: Any diagnosed kidney conditions
* Cardiovascular Disease: Any diagnosed cardiovascular conditions
* Hypertension: Diagnosed high blood pressure
* Recent Illness or Infection: Any illness or infection within the past 30 days that could affect study outcomes
* Tobacco or Nicotine Use: Current use of tobacco or nicotine products (e.g., smoking, vaping)
* Phenylketonuria (PKU): A genetic disorder affecting phenylalanine metabolism, due to the presence of aspartame in Diet Coke
* Medication Use: Use of medications or supplements that affect glucose metabolism, insulin response, or appetite
* Intermittent Fasting: Engagement in intermittent fasting or inconsistent time-restricted feeding patterns
* Other Health Conditions: Any other health conditions that, in the opinion of the investigators, could interfere with study participation or outcomes

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological males only
Enrollment: 10 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Glucose | At baseline and at 15, 30, 60, 90, and 120 minutes
  The AUC of plasma glucose concentrations will be compared between the four conditions.
Satiety | At baseline and at 15, 30, 60, 90, and 120 minutes
  Subjective feelings of hunger and fullness following beverage consumption will be measured using a self-created 10-point Likert-type scale in which higher numbers will mean higher satiety/fullness. Minimum score, equal to zero, means extremely hungry, whereas maximum score, equal to 10, means extremely stuffed.
Insulin | At baseline and at 15, 30, 60, 90, and 120 minutes
  The AUC of plasma insulin concentrations will be compared between the 4 conditions.
GLP-1 | At baseline and at 15, 30, 60, 90, and 120 minutes
  The AUC of GLP-1 will be compared between the 4 conditions.

SECONDARY OUTCOMES:
Gastrointestinal Symptoms | 24h after each the visit
  Participants will fill out our self-created GI Symptoms Questionnaire to report the severity of any of the following GI symptoms: bloating, gas, stomach pain, nausea, diarrhea, constipation, urgency to use the restroom, and any other symptoms. Severity will be measured on a scale of 0 to 10, where 0 means none and 10 means severe/unbearable. If any symptoms are present, they will then be asked to report their timing with regards to drink consumption (N/A, <15 min, 15-30 min, 30-60 min, 60-120 min, and >120 min). Participants will also be asked to write down the length of this symptomatology (N/A, <30 min, 30-60 min, 1-3 h, >3h, and symptoms still ongoing). A comparison between the 4 conditions will be performed.
Beverage Palatability | After beverage consumption
  Participants will fill out a self-created Beverage Rating Questionnaire in which they will grade the drink's taste, sweetness, aftertaste, texture, and carbonation of the drink by using a Likert-scale 0-10 in which 0 means "Completely absent or extreme in an unpleasant way" and 10 means "Outstanding, ideal, enhances the experience". Participants will also be asked to report their overall beverage satisfaction by using from 5 options going from 0= None at all to 5= A great deal. Lastly, participants will be asked to compare the consumed drink (blinded) to other drinks he has drunk in the past and report if the current drink was not better or worse (NA), much worse, womewhat worse, about the same, somewhat better, or much better compared to Olipop, Poppi, Diet Coke, and Coca Cola. Comparison between the four conditions will be performed.

OTHER OUTCOMES:
Body Composition | At the baseline of visit 2.
  DEXA scans will be used to measure total fat mass, total lean mass, bone mineral density, and visceral adipose tissue.
Fasting capillary glucose | At the baseline of visit 1
  A single finger-stick will be collected at the beginning of the first visit to confirm eligibility. A glucose value of <100 mg/dl is needed to enroll in the study.
Fasting capillary HbA1C | At the baseline of visit 1
  A single finger stick will be collected to corroborate eligibility at the beginning of the first visit. A value of HbA1C <6.5% is required to enroll in the study.
Blood pressure | Baseline
  Systolic and diastolic blood pressure will be measured at the beginning of each visit using a digital blood pressure cuff (SBP >180 mmHg or DBP >110 mmHg prompts unenrollment and referral to a healthcare provider). Comparison between the four conditions will be performed.
Dietary habits | Baseline of visit 1
  A 3-day food log (2 weekdays and 1 weekend) will be applied to participants during visit 1. The objective of this analysis is to provide baseline data to assess for dietary influences on metabolic outcomes.
Non-Caloric Sweetener Questionnaire | Baseline of visit 1
  Participants will fill out a long, self-created Artificial Sweetener Intake Questionnaire in which participants will be asked about the amount (8 oz, 12 oz, 16 oz, and >20 oz) and frequency (never, 1x/week, 2-3x/week, 4-6x/week, 1x/day, 2x/day, >3x/day) at which dietary products that contain non-caloric sweeteners are consumed. Foods include different brands of flavored waters, juices, soft drinks, teas, chocolate drinks, coffee drinks, sweeteners, coffee creamer, energy drinks, protein drinks, pre-workouts, yogurts, ice creams, cookies, bars, candy, jello, pudding, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Additional analyses may be conducted on our data following the conclusion of this study. However, if the study and the analyses described herein are completed and no further analyses are planned by our research team, the data may be made available upon request by contacting Elisa Marroquín

REFERENCES:
- [Background] Steinert RE, Frey F, Topfer A, Drewe J, Beglinger C. Effects of carbohydrate sugars and artificial sweeteners on appetite and the secretion of gastrointestinal satiety peptides. Br J Nutr. 2011 May;105(9):1320-8. doi: 10.1017/S000711451000512X. Epub 2011 Jan 24. PMID 21255472
- [Background] Brown RJ, Walter M, Rother KI. Ingestion of diet soda before a glucose load augments glucagon-like peptide-1 secretion. Diabetes Care. 2009 Dec;32(12):2184-6. doi: 10.2337/dc09-1185. Epub 2009 Oct 6. PMID 19808921
- [Background] Kim Y, Keogh JB, Clifton PM. Consumption of a Beverage Containing Aspartame and Acesulfame K for Two Weeks Does Not Adversely Influence Glucose Metabolism in Adult Males and Females: A Randomized Crossover Study. Int J Environ Res Public Health. 2020 Dec 4;17(23):9049. doi: 10.3390/ijerph17239049. PMID 33291649
- [Background] Bian X, Chi L, Gao B, Tu P, Ru H, Lu K. The artificial sweetener acesulfame potassium affects the gut microbiome and body weight gain in CD-1 mice. PLoS One. 2017 Jun 8;12(6):e0178426. doi: 10.1371/journal.pone.0178426. eCollection 2017. PMID 28594855
- [Background] Ahmad SY, Friel JK, Mackay DS. Effect of sucralose and aspartame on glucose metabolism and gut hormones. Nutr Rev. 2020 Sep 1;78(9):725-746. doi: 10.1093/nutrit/nuz099. PMID 32065635
- [Background] Vandeputte D, Falony G, Vieira-Silva S, Wang J, Sailer M, Theis S, Verbeke K, Raes J. Prebiotic inulin-type fructans induce specific changes in the human gut microbiota. Gut. 2017 Nov;66(11):1968-1974. doi: 10.1136/gutjnl-2016-313271. Epub 2017 Feb 17. PMID 28213610
- [Background] Cani PD, Lecourt E, Dewulf EM, Sohet FM, Pachikian BD, Naslain D, De Backer F, Neyrinck AM, Delzenne NM. Gut microbiota fermentation of prebiotics increases satietogenic and incretin gut peptide production with consequences for appetite sensation and glucose response after a meal. Am J Clin Nutr. 2009 Nov;90(5):1236-43. doi: 10.3945/ajcn.2009.28095. Epub 2009 Sep 23. PMID 19776140